CLINICAL TRIAL: NCT05919147
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Neuroendocrine Effects of Pioglitazone in Patients With Cancer and Cachexia
Brief Title: The Neuroendocrine Effects of Pioglitazone in Patients With Cancer and Cachexia
Acronym: TRACE-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Steven Heymsfield, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PBRC 2023-013
Record Dates: First submitted 2023-06-12; First posted 2023-06-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone 45 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone 45 mg — The dose of pioglitazone will not exceed 45 mg once daily. Pioglitazone dose will titrate progressively over the first three weeks.
  Arms: Pioglitazone
Drug: Placebo — Placebo will have the same appearance as the active drug.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is evaluate the effect of pioglitazone compared with placebo on skeletal muscle insulin sensitivity in subjects with cancer and cachexia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented histologic or cytologic diagnosis of non-small-cell lung cancer or gastrointestinal cancer that is locally advanced and inoperable or metastatic (e.g., spread to distant organs)
* Cachexia defined by Fearon criteria
* Insulin resistance syndrome, defined with the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
* Ability to provide written informed consent, willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures
* Provide written approval by a qualified healthcare professional
* Allow the collection and storage of biospecimens and data for future use

Exclusion Criteria:

* Prior diagnosis of type 2 diabetes
* Prior or current thiazolidinedione (TZD) therapy
* Known hypersensitivity to TZD
* New York Heart Association (NYHA) class I-IV heart failure
* History of or actively treated bladder cancer
* Current use of CYP2C inhibitor (e.g., gemfibrozil) or CYP2C inducer (e.g., rifampin)
* Inadequate hepatic function
* Currently pregnant, breastfeeding, or planning to become pregnant within the next 16 weeks
* Contraindications to magnetic resonance imaging (e.g., implanted cardiac device, cochlear implant)
* Any other condition that, in the investigator's opinion, would preclude participation or successful compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle insulin sensitivity | Baseline, Week 12
  Quantified using hyperinsulinemic-euglycemic clamp

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes